CLINICAL TRIAL: NCT04375176
Title: Study of Immune-mediated Mechanisms in Patients Tested Positive for SARS-CoV-2: Phenotypic and Functional Analysis of Monocytes and NK Cells in the Blood of Subjects Affected by Covid 19
Brief Title: Monocytes and NK Cells Activity in Covid-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Ietto Giuseppe, Adjunct Professor, M.D., Università degli Studi dell'Insubria
Other Study IDs: 67/2020
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome Coronavirus 2; Immunomodulation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood sample (15 mL in EDTA solution test tube).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tested positive for SARS-CoV-2: Patients, tested positive for SARS-CoV-2, will be recruited in E.R. of the "Ospedale Di Circolo - ASST Settelaghi" Teaching Hospital in Varese.
  Interventions: Diagnostic Test: Study of immune-mediated mechanisms in patients tested positive for SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Study of immune-mediated mechanisms in patients tested positive for SARS-CoV-2 — Phenotypic and functional analysis of monocytes and NK cells

SUMMARY:
SARS-CoV-2 belong to beta-coronavirus family and its transmission route and symptoms follow those of all community-acquired coronaviruses. The main difference of the novel Coronavirus is the higher mortality rate, that is around 3%.

Death rate is over 1% only for patients over 50 years old, whereas until 40 years old is under 0,4%. No fatalities are declared among children under 10 years old to date. Death rate is almost double for male rather than female. This distribution of mortality rate according to age of infected patients could be only partially ascribed to other comorbidities in addition to great age. In fact, patients with no pre-existing conditions have however a case fatality rate of 0,9%.

The almost null rate of severe illness in children and generally in patients younger than 40 years old is quite un-explicable. Infant, children and young people could be infected but infection is rapidly self-limited or without symptoms. Older patients undergo severe lung injury as consequence of an immune response that is late in coming.

Possible explanation of these phenomena could be something, which assure ability to prompt response to SARS-CoV-2 in younger people independently from the novelty of the virus itself.

It would seem to be that younger people are already sensitized to the antigens of the virus without a previous contact.

This immunity is not really specific, but "partially specific" for many antigens of the virus, however able to limit the infection in the organism. Something stimulated the immune system and it scattered immunity against more and more antigens present. Children are the age group mostly exposed to all community-circulating viruses.

This immunity is not persistent but progressively fade out. It protects from the age of two, when the hypothetical stimulation occurs, to the fifth decade because of its slow decrease.

The only external stimulation, which healthy people receive are vaccines. All vaccinations and especially tetanic, diphtheria toxoids and inactivated bacteria as pertussis could stimulate immune system. They develop the specific immunity but generate also a sprouting immunity against antigens in transit, as coronaviruses and other community-circulating viruses.

The developed immunity gives some protection against multiple viral infection for years until the natural fade out.

After the fifth decade, that immunity is slower to be recall and reactivated. Additionally, transplant recipients and HIV infected patients, which have an immune system inhibited, unexpectedly, do not seem to suffer the worst complications of SARS-CoV-2 infection. An immune system imbalance could be play a pivotal role during the reaction to the virus, limiting destructive consequences of excessive inflammation.

According to the medical hypothesis on which the protocol is based on, young people could benefit from a functional adaptation of innate immune cells induced through epigenetic reprogramming and, especially, a pre-existing "partially specific" immunity to the community viruses caused by "bystander effect" of preceding vaccinations. In this study, we will explore the main differences existing among patients infected by SARS-CoV-2 who experience the illness at different degree of severity. We suppose to recognize different populations of patients, each one with a specific immunological pattern. It could differ in terms of cytokines, soluble factors serum level and immune cells activity both of the innate compartment and of the acquired one. The proof of a role of these immunological phenomena in the pathogenesis of Covid-19 are bases for implementation of therapeutic immunomodulatory treatments. In addition, the definition of an immunological risk profile could tailor established therapies to each kind of patient.

DETAILED DESCRIPTION:
According to the medical hypothesis on which the protocol is based on, young people could benefit from a functional adaptation of innate immune cells induced through epigenetic reprogramming and, especially, a pre-existing "partially specific" immunity to the community viruses caused by "bystander effect" of preceding vaccinations. In this study, we will explore the main differences existing among patients infected by SARS-CoV-2 who experience the illness at different degree of severity. We suppose to recognize different populations of patients, each one with a specific immunological pattern. It could differ in terms of cytokines, soluble factors serum level and immune cells activity both of the innate compartment and of the acquired one.

Data will be collected using 3 approaches:

* An experimental analysis, for clusters of patients, to study the innate immune response and to identify the genetic profiles.
* An epidemiological analysis, in order to identify the patients' vaccination history;
* A clinical analysis, to detect the immunological profile;

For the specific analysis, to study the innate immune response and to identify the genetic profiles, scientists will analyze, from the peripheral blood, NK cells, monocytes, CD4 and CD8 T cells of both groups: healthy patients (tested negative for SARS-CoV-2) and sick patients of the subgroups (AS 19, PAU19, POL19, ARD19).

From different groups of patients, blood samples (10-15 mL) will be drawn into EDTA tubes, centrifuged at 360 g for 10 minutes to obtain plasma that it will be stored at -80°C for subsequent analysis for cytokines and chemokines of interest by ELISA (IL-1b, IL-6, TNF, IFN-a, IL-10, IL-12, CCL2 and CXCL10) at the end of enrolment.

The cell pellets will be brought back to the initial volume with PBS and diluted 1:1 (v/v), and then subjected to a density gradient stratification with Ficoll Histopaque-1077, at 500 g for 30 minutes. The Peripheral Blood Mononuclear Cells (PBMCs) derived from the white ring will be collected, washed twice in PBS, and then used for subsequent experiments using a flow cytometer assay (REFF). The in vitro culture using PBMCs can vary from ex vivo 1 day to a few days, and cells will be maintained in RPMI 1640 medium, supplemented with 10% fetal bovine serum (FBS), 2 mM l-glutamine, 100 U/mL penicillin and 100 μg/mL streptomycin (P/S), at 37°C, 5% CO2.

To perform ex vivo fluorescence-activated cell sorter (FACS) phenotype analysis, 2.5x105 of fresh total PBMCs per FACS tube will be stained for 30 minutes at 4°C with monoclonal antibodies (mAbs) as follows: CD3-PerCP, CD56-APC, CD16-FITC, NKG2A-PE, NKG2C-PE, NKGD2-PE, DNAM-1-PE, CD25-PE, CD69-PE. Following Forward/Side Scatter setting, NK cells will be identified into two cell subsets, i.e. as CD3- and CD56dim CD16+ cells (CD56dim NK cells, the major subset, about 90%), and CD3- and CD56bright CD16-/low cells (CD56bright NK cells, the minor subset, about 10%). Other markers expression will be evaluated on both subsets of gated cells.

For ex vivo FACS evaluation of monocytes phenotype analysis, 2.5x105 of fresh total PBMCs per FACS tube will be stained for 30 minutes at 4°C with mAbs as follows: CD45-APC, CD14-FITC and CD16-V450, PE-CD209, PE-CD80. Following Forward/Side Scatter setting, monocytes will be identified into three subsets, i.e. as CD14+ and CD16- cells (the main subset, about 90%), CD14+ CD16+ (the minor subset, about 10%), and CD14-/low CD16+ (the other minor subset).

We will also evaluate phenotype for CD4 and CD8 T cells and CD4/CD8 T ratio using 2x105 of fresh total PBMCs, as previously described, with following mAbs: CD3-PerCP, CD4-APC, CD8-V450 as well as T regulatory (Treg) cells, as CD3-PerCP, CD4-APC, CD25-PE.

PBMCs will be also in vitro stimulated for 4 h with different types of stimuli, such as LPS (recognized by the TLR4), poly(I:C) (recognized by the TLR3), poly (I:C) plus IL-2 plus IL-12, and phorbol myristate acetate (PMA) plus ionomycin in presence of monensin and brefeldin. This procedure will allow studying specific cytokine/chemokine production from NK cells and monocytes by using a FACS intracellular assay, as described previously (REFF). For NK cells, we will measure IFN-a-PE, TNF-PE, CCL2-PE, CXCL10-PE and CD107a-PE (degranulation marker). For monocytes we will investigate: IL-6-PE, TNFa-PE, IL-12-PE, CXCL10-PE (M1-type pro-inflammatory markers) and TGFb-PE, IL-10-PE, CCL18-PE (M2-type anti-inflammatory markers) Whenever the quantity of PBMCs is sufficient, other functional in vitro tests on NK cells and monocytes will be set up. In particular, PBMCs will be studied for 4 h NK cell degranulation/cytotoxic function towards erytroleucemic K562 cell line assessing surface CD107a-PE using a flow cytofluorimetric assay (REFF).

Whenever the quantity of PBMCs is sufficient, monocytes will be purified using anti-CD14 microbeads with magnetic separator and NK cells with RosetteSep kit to obtain >90% purified cell populations.

Purified monocytes and purified NK could be maintained separated or together in culture using RPMI 1640 medium with 10%FBS, and supplemented with M-CSF and IL-2, respectively, stimulated with different stimuli (see above), and then checked for intracellular cytokines/chemokines of interest (see above). At the same time the supernatants (conditioned medium, CM) could be harvested at the end of in vitro incubation culture and assessed for cytokines/chemokines using ELISA (IL-1b, IL-6, TNFa, IFNa, IL-10, IL-12, CXCL10).

The 4-5 days in vitro culture of monocytes will be further stimulated 24 h with LPS plus IFNg (M1 stimulus) or (IL-4) (M2 stimulus) to investigate macrophage polarization studying surface M1 markers (TNF, CXCL10) or M2 markers (IL-10, CCL18) to check the prevalence of macrophage polarization in different groups of Covid-19 patients.

The epidemiological analysis will be carried out integrating both vaccination history and the data daily collected after hospital admission. ATS Insubria archives will provides missing data.

Considering the immunological profile, patients with Covid-19 will be tested for routine examinations and the following:

* lymphocyte immunophenotyping;
* determination of C3 and C4 complement fractions activity;
* immunoglobulin (IgG, IgM, IgA, IgE) serum level;
* serum protein electrophoresis;
* Angiotensin Converting Enzyme (ACE) serum level;
* CMV (Citomegalovirus) serology test;
* IL-6 serum level.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18
* SARS-CoV-2 documented infection

Exclusion Criteria:

* Refusal to the sign the agreement (informed consent);
* Inability to sign the agreement;
* HIV, HCV, HBV (positive to HBsAg) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients tested positive for SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Immune cells activity | 6 months
  Scientists' hypothesis is that monocytes, NK, CD4 AND CD8 T cells, in patients with severe infection to SARS-CoV-2, show an impairment in their function: cells reveal an overpowering hyperactivity that provokes a pathologic inflammatory response with a massive production of proinflammatory cytokine, edema and pulmonary fibrosis.

SECONDARY OUTCOMES:
Protective factors and new therapeutic strategies | 6 months
  The secondary objectives are to correlate clinical data and vaccination history with laboratory immune pattern to identify protective factors for Covid 19 and open paths for new therapeutic strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Carcano, Professor, Study Chair — Università degli Studi dell'Insubria; Giuseppe Ietto, M.D., Principal Investigator — Università degli Studi dell'Insubria; Lorenzo Mortara, Professor, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- ATS Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ietto G. SARS - CoV-2: Reasons of epidemiology of severe ill disease cases and therapeutic approach using trivalent vaccine (tetanus, diphtheria and Bordetella pertussis). Med Hypotheses. 2020 Aug;141:109779. doi: 10.1016/j.mehy.2020.109779. Epub 2020 Apr 22. PMID 32387756
- [Background] Netea MG, Dominguez-Andres J, Barreiro LB, Chavakis T, Divangahi M, Fuchs E, Joosten LAB, van der Meer JWM, Mhlanga MM, Mulder WJM, Riksen NP, Schlitzer A, Schultze JL, Stabell Benn C, Sun JC, Xavier RJ, Latz E. Defining trained immunity and its role in health and disease. Nat Rev Immunol. 2020 Jun;20(6):375-388. doi: 10.1038/s41577-020-0285-6. Epub 2020 Mar 4. PMID 32132681
- [Background] Murray PJ, Allen JE, Biswas SK, Fisher EA, Gilroy DW, Goerdt S, Gordon S, Hamilton JA, Ivashkiv LB, Lawrence T, Locati M, Mantovani A, Martinez FO, Mege JL, Mosser DM, Natoli G, Saeij JP, Schultze JL, Shirey KA, Sica A, Suttles J, Udalova I, van Ginderachter JA, Vogel SN, Wynn TA. Macrophage activation and polarization: nomenclature and experimental guidelines. Immunity. 2014 Jul 17;41(1):14-20. doi: 10.1016/j.immuni.2014.06.008. PMID 25035950
- [Background] Noonan DM, De Lerma Barbaro A, Vannini N, Mortara L, Albini A. Inflammation, inflammatory cells and angiogenesis: decisions and indecisions. Cancer Metastasis Rev. 2008 Mar;27(1):31-40. doi: 10.1007/s10555-007-9108-5. PMID 18087678
- [Background] Parisi L, Gini E, Baci D, Tremolati M, Fanuli M, Bassani B, Farronato G, Bruno A, Mortara L. Macrophage Polarization in Chronic Inflammatory Diseases: Killers or Builders? J Immunol Res. 2018 Jan 14;2018:8917804. doi: 10.1155/2018/8917804. eCollection 2018. PMID 29507865
- [Background] Benn CS, Netea MG, Selin LK, Aaby P. A small jab - a big effect: nonspecific immunomodulation by vaccines. Trends Immunol. 2013 Sep;34(9):431-9. doi: 10.1016/j.it.2013.04.004. Epub 2013 May 14. PMID 23680130
- [Background] Bruno A, Focaccetti C, Pagani A, Imperatori AS, Spagnoletti M, Rotolo N, Cantelmo AR, Franzi F, Capella C, Ferlazzo G, Mortara L, Albini A, Noonan DM. The proangiogenic phenotype of natural killer cells in patients with non-small cell lung cancer. Neoplasia. 2013 Feb;15(2):133-42. doi: 10.1593/neo.121758. PMID 23441128
- [Background] Bruno A, Bassani B, D'Urso DG, Pitaku I, Cassinotti E, Pelosi G, Boni L, Dominioni L, Noonan DM, Mortara L, Albini A. Angiogenin and the MMP9-TIMP2 axis are up-regulated in proangiogenic, decidual NK-like cells from patients with colorectal cancer. FASEB J. 2018 Oct;32(10):5365-5377. doi: 10.1096/fj.201701103R. Epub 2018 May 15. PMID 29763380
- [Background] Bassani B, Baci D, Gallazzi M, Poggi A, Bruno A, Mortara L. Natural Killer Cells as Key Players of Tumor Progression and Angiogenesis: Old and Novel Tools to Divert Their Pro-Tumor Activities into Potent Anti-Tumor Effects. Cancers (Basel). 2019 Apr 1;11(4):461. doi: 10.3390/cancers11040461. PMID 30939820
- [Background] Morandi F, Horenstein AL, Chillemi A, Quarona V, Chiesa S, Imperatori A, Zanellato S, Mortara L, Gattorno M, Pistoia V, Malavasi F. CD56brightCD16- NK Cells Produce Adenosine through a CD38-Mediated Pathway and Act as Regulatory Cells Inhibiting Autologous CD4+ T Cell Proliferation. J Immunol. 2015 Aug 1;195(3):965-72. doi: 10.4049/jimmunol.1500591. Epub 2015 Jun 19. PMID 26091716
- [Derived] Ietto G, Mortara L, Dalla Gasperina D, Iovino D, Azzi L, Baj A, Ageno W, Genoni AP, Acquati F, Gallazzi M, Spina G, Coco G, Pierin F, Noonan D, Vigezzi A, Monti E, Iori V, Masci F, Franchi C, Di Saverio S, Carcano G. Immune-Mediated Mechanisms in Patients Testing Positive for SARS-CoV-2: Protocol for a Multianalysis Study. JMIR Res Protoc. 2022 Jan 25;11(1):e29892. doi: 10.2196/29892. PMID 34854818